CLINICAL TRIAL: NCT04133129
Title: Study of the Effects of a Structured Training Program on People at Risk of Developing Metabolic Syndrome
Brief Title: Effects of HIIT on Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Coventry University (Other)
Collaborators: INGESPORT HEALTH AND SPA CONSULTING SL (Unknown)
Responsible Party: Principal Investigator, Ismael Serrablo, Principle Investigator, Coventry University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P72554
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Dyslipidemias; Metabolic Syndrome; Sedentary Behavior; Obesity; Blood Pressure
Keywords: HIIT; High Intensity Interval Training; Medium Intensity Continuous Training; Interval Training; Exercise; Physical Activity; Exercise Training
MeSH Terms: conditions — Dyslipidemias; Metabolic Syndrome; Sedentary Behavior; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are only assigned to one of 3 possible groups for the duration of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LV-High Intensity Interval Training (Experimental): 2 x 4 minutes at 85%-95% of Heart rate max.
  Interventions: Behavioral: Low Volume-High Intensity Interval Training
- Moderate Intensity Continuous Training (Experimental): 1 x 45 minutes at 65%-75% of Heart rate max.
  Interventions: Behavioral: Moderate Intensity Continuous Training
- Control Group (No Intervention): They will not be prescribed any training and will be asked to continue with their normal lifestyle.

INTERVENTIONS:
Behavioral: Low Volume-High Intensity Interval Training — On a treadmill, a 2 minute warm-up will be followed by 2 bouts of 4 minutes at an intensity between 85% and 95% of Maximum Heart Rate (HRmax) interspersed by a 2 minutes recovery bout at 70% of heart rate max, followed by a 3 minutes Cool Down
  Other Names: HIIT; LV-HIIT
  Arms: LV-High Intensity Interval Training
Behavioral: Moderate Intensity Continuous Training — On a treadmill,a 2-minute warm-up will be followed by 45 minutes at 65%-75% of Heart Rate max followed by 3 minutes cool down.
  Other Names: MICT
  Arms: Moderate Intensity Continuous Training

SUMMARY:
The project aims to find out the differences between two different types of structured training interventions have on the lipid profile of persons with diagnosed dyslipidemia. Each training intervention will last for 12 weeks. Subjects participating in the project will undergo a series of tests before and after the training intervention which will allow us to make conclusions.

DETAILED DESCRIPTION:
The purpose of this project is to compare the effect that two different types of aerobic training modes have on the lipid profile of subjects with pre-symptoms of metabolic syndrome. One training mode will involve High-Intensity Interval Training and the other will involve medium intensity continuous training. The desired outcomes of this project are to know the effects of both modes of training have on the long-term on the lipid profile in order to help develop a nonpharmacologic alternative to prevent or treat metabolic syndrome and to know how affective and enjoyment responses are affected by the different modes of training. The Project lasts for 16 weeks. Training will take place during weeks 3 and 14 of the project. The project will be described fully to the participants during the 1st week. In addition to this, their rights as participants will be explained in addition to any possible ethical issues that might require clarifying. Once the subjects have agreed to take part in the research they will undergo a series of tests in order to asses their cardiorespiratory fitness and their lipids profile. Before starting the training intervention participants will be randomly assigned to one of the 3 different groups; Control, Medium Intensity Continuous Training and Low Volume High-Intensity Interval Training. Between weeks 3 and 14 subjects will take part in 3 training sessions per week. At week 15 and 16 subjects will undergo the same tests as during week 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Fasted Blood Glucose >100 mg/dL
* Total Cholesterol >200 mg/dL
* Blood Pressure >130/90 mmHg
* Do not partake in more than 150 min/week of moderate to vigorous exercise

Exclusion Criteria:

* Existing or past medical history of vascular disease, cancer, diabetes, osteoporosis, neurological, kidney, pulmonary, digestive (Coeliac disease), thyroidal disease.
* Musculoskeletal injuries
* Neuromuscular disorders or injuries
* Individuals with a pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-03-02 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical: Lipid Profile | 0 to 12 weeks
  Evaluate change in Very Low-Density Lipoproteins (VLDL), High Density Lipoprotein (HDL), and Low-Density Lipoprotein (LDL) in (mg/dl) with Liposcale® test, an advanced lipoprotein test based on 2D Nuclear Magnetic Resonance (NMR).
Blood Pressure (mmHg) | 0 to 12 weeks
  Evaluate change in Systolic and Diastolic Blood Pressure
Cardiorespiratory Fitness (ml/kg/min) | 0 to 12 weeks
  Evaluate change in maximal oxygen uptake (VO2max) via breath by breath analysis performed on a treadmill.
Changes in Body Composition (kg) | 0 to 12 weeks
  Evaluate changes in Fat-free mass, fat mass, skeletal muscle mass measured by bio-electrical impedance analysis.

SECONDARY OUTCOMES:
Changes in exercise enjoyment | 0 to 12 weeks
  The investigators will assess perceived exercise enjoyment at baseline and post intervention using The Physical Activity Enjoyment Scale (PACES). (PACES) is an 18-item measure, scored on a 7-point bipolar scale based on the instruction; "Please rate how you feel at the moment about the physical activity you have been doing:"
Change in Behavioural Regulations in Exercise Questionnaire-2 (BREQ-2) over time | 0 to 12 weeks
  Behavioural Regulations in Exercise Questionnaire-2 (BREQ-2) is a 19 item self-report scale. It uses a Likert-type scale of 5 points, where 0 = not true for me and 4 = very true for me

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Horton, PhD, Study Director — Coventry University; Alfonso Jimenez, PhD, Study Director — GOfit and Sheffield Hallam University; Ismael Serrablo, MSc, Principal Investigator — Coventry University
Locations (1):
- CDM GO fit Vallehermoso, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No